CLINICAL TRIAL: NCT04635774
Title: Intranasal Insulin and Neurocognitive Function
Brief Title: Post Operative Delirium Study
Acronym: PODS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Participants were unable to be enrolled
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Frank E Weinhold Pharm.D., M.S., Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00146489
Record Dates: First submitted 2020-11-06; First posted 2020-11-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Delirium
Keywords: Insulin
MeSH Terms: conditions — Delirium; Insulin Resistance | interventions — Insulin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is double-blind, randomized, placebo controlled. Neither the physician, patient, nor investigator will be aware of which patient is receiving insulin and which is receiving placebo. The treatment group will receive 40 IU via four activations of an intranasal spray. The placebo group will receive four activations of an intranasal spray containing placebo (normal saline).
  Both groups of patients receiving the insulin or placebo as intervention will be assessed with the CAM assessment at 10 min, 30min, and 60 min, and 6hr.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigational pharmacist will use randomization software to randomize numbers 1-30. Each number will be randomized to either active drug (regular insulin) or placebo (normal saline).The investigational pharmacist will have the randomization table should un-blinding be required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Active Comparator): The treatment group will receive 40 IU via four activations of an intranasal spray.
  Interventions: Drug: Insulin
- Placebo Group (Placebo Comparator): The placebo group will receive four activations of an intranasal spray containing placebo (normal saline).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Insulin — 40 IU via four activations of an intranasal spray
  Arms: Treatment Group
Drug: Saline — Four activations of an intranasal spray containing placebo (normal saline).
  Arms: Placebo Group

SUMMARY:
Post-operative delirium happens when patients wake up from anesthesia. Patients experiencing post-operative delirium are very confused, not being able to think or function "normally". These patients are hard to take care of and they tend to have more dementia as they age compared to patients who don't experience post-operative delirium. Intranasal insulin has been shown to reverse confusion associated with Alzheimer's disease (humans) and AIDS (mice).

Intranasal insulin has been safely administered to 1092 patients in 38 different studies. There were no cases of clinically low blood sugar and a few cases of mild nasal irritation that happened also with salt water when the subjects received multiple intranasal doses.

No one has tried to reverse post-operative delirium with intranasal insulin. The delirium associated with Alzheimer's Disease and AIDS have very similar symptoms and what happens in the brain is very similar also.

The investigators intent is to administer intranasal insulin to patients exhibiting post-operative delirium in order to reverse the symptoms because the investigators think that the three disease states are closely related and intranasal insulin has had some success in reversing the delirium in the other two disease states.

ELIGIBILITY:
Inclusion Criteria:

* All patients (>65 years of age) undergoing elective surgery using vapor anesthesia displaying post-operative delirium as defined by a CAM evaluation within time to PACU discharge post-surgery are eligible.
* Those patients 65 and older undergoing surgery using vapor anesthesia, who are consented but do not exhibit delirium and are not part of the study are still considered recruited subjects, but are not in the active study.

Exclusion Criteria:

* Patients with a history of severe dementia, anoxic brain injury, or neuromuscular disorders
* Non-English-speaking patients
* Planned use of drugs that effect plasma glucose concentration during the first four hours of surgery
* thiazolidinediones
* hormones which may affect plasma glucose or insulin
* contraceptive, diphenylhydantoin
* patients with allergy to insulin
* acromegaly
* Cushing's syndrome
* hyperthyroidism and pheochromocytoma
* renal impairment
* pregnant and lactating women
* base line blood glucose < 3.9 mmol/L

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of intranasal insulin in resolving post-operative delirium | 10 min post diagnosis
  Measured by administering the Confusion Assessment Method (CAM) tool
Efficacy of intranasal insulin in resolving post-operative delirium | 30 min post diagnosis
  Measured by administering the Confusion Assessment Method tool
Efficacy of intranasal insulin in resolving post-operative delirium | 60 min post diagnosis
  Measured by administering the Confusion Assessment Method tool
Efficacy of intranasal insulin in resolving post-operative delirium | 6 hours post diagnosis
  Measured by administering the Confusion Assessment Method tool

SECONDARY OUTCOMES:
Length of stay in the post-anesthesia care unit (PACU) | Time from admission to the PACU until discharge from PACU, up to 18 hours from admission to the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Frank Weinhold, Pharm.D., MS, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No